CLINICAL TRIAL: NCT03223051
Title: Development of a Space Exploration Assessment for Children With Spinal Muscular Atrophy
Acronym: ExplorASI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre d'Investigation Clinique et Technologique 805 (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2017-A01017-46
Record Dates: First submitted 2017-07-18; First posted 2017-07-19 (Actual); Last update posted 2019-11-25 (Actual); Status verified 2019-11

CONDITIONS: Spinal Muscular Atrophy; Assessment, Self
Keywords: Spinal Muscular Atrophy; Children; Motor assessment; Space exploration; Upper limbs
MeSH Terms: conditions — Muscular Atrophy, Spinal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Evaluation (Experimental): Included patients will be invited to participate in 1 session, to be evaluated with the Motor Function Measure and the new test of space exploration, during 2 hours maximum, to compare scores with these 2 tests.
  An occupational therapist will be required to install the patient in front of the table and to give the instructions.
  Interventions: Other: Motor assessment

INTERVENTIONS:
Other: Motor assessment — An occupational therapist install the patient sitting in front of the test board and tell him the instructions

SUMMARY:
The aim of this randomized study is to develop a new motor assessment of space exploration in a 2D environment with upper limbs for children with spinal muscular atrophy 1 and 2 from 3 until 16 years old.

DETAILED DESCRIPTION:
Thirty children are included in the prospective randomized study. They are evaluated with the new test, Space Exploration Test (TES), and with the Motor Function Measure (MFM), a gold standard scale. The objective is to compare the results and to demonstrate the complementarity of the two tools.

ELIGIBILITY:
Inclusion Criteria:

* children, girls and boys, from 3 to 16 years old,
* with Spinal Motor Atrophy 1 and 2
* with social protection

Exclusion Criteria:

* cognitive disorders preventing understanding

Ages: 3 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2017-09-07 (Actual); Primary Completion 2019-11-22 (Actual); Study Completion 2019-11-22 (Actual)

PRIMARY OUTCOMES:
Motor Function Measure (MFM) | 1 hour
  Clinical Evaluation

SECONDARY OUTCOMES:
Space Exploration Test (SET) | 20 minutes
  The SET is made through a test board 170 cm long and 60 cm deep, developed by in our lab

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas ROCHE, MDphD, Principal Investigator — Raymond Poincare HOSPITAL
Locations (2):
- France (2):
  - Hopital Raymond Poincare, Garches
  - Nicolas ROCHE, Md PhD, Garches

IPD SHARING:
Plan to Share IPD: No